CLINICAL TRIAL: NCT01966055
Title: A Phase 1, Open-label, Multi-center Study to Determine the PK and Safety of Solithromycin as Add-on Therapy in Adolescents With Suspected or Confirmed Bacterial Infection
Brief Title: Pharmacokinetics and Safety of Solithromycin Capsules in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE01-119
Record Dates: First submitted 2013-10-15; First posted 2013-10-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — solithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Solithromycin (Experimental)
  Interventions: Drug: Solithromycin

INTERVENTIONS:
Drug: Solithromycin

SUMMARY:
A study of the safety and pharmacokinetics of solithromycin capsules in adolescents

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 yo male or female with suspected or confirmed bacterial infection

Exclusion Criteria:

* Bacterial meningitis
* Clinical significant concomitant medical condition

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of solithromycin in adolescents | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen-Wolkowiez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (11):
- United States (11):
  - Little Rock, Arkansas
  - San Diego, California
  - Chicago, Illinois
  - Louisville, Kentucky
  - Ann Arbor, Michigan
  - Hackensack, New Jersey
  - New York, New York
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Galveston, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Beechinor RJ, Cohen-Wolkowiez M, Jasion T, Hornik CP, Lang JE, Hernandez R, Gonzalez D. A Dried Blood Spot Analysis for Solithromycin in Adolescents, Children, and Infants: A Short Communication. Ther Drug Monit. 2019 Dec;41(6):761-765. doi: 10.1097/FTD.0000000000000670. PMID 31318840
- [Derived] Gonzalez D, James LP, Al-Uzri A, Bosheva M, Adler-Shohet FC, Mendley SR, Bradley JS, Espinosa C, Tsonkova E, Moffett K, Marquez L, Simonsen KA, Stoilov S, Boakye-Agyeman F, Jasion T, Hornik CP, Hernandez R, Benjamin DK Jr, Cohen-Wolkowiez M. Population Pharmacokinetics and Safety of Solithromycin following Intravenous and Oral Administration in Infants, Children, and Adolescents. Antimicrob Agents Chemother. 2018 Jul 27;62(8):e00692-18. doi: 10.1128/AAC.00692-18. Print 2018 Aug. PMID 29891609
- [Derived] Gonzalez D, Palazzi DL, Bhattacharya-Mithal L, Al-Uzri A, James LP, Bradley J, Neu N, Jasion T, Hornik CP, Smith PB, Benjamin DK Jr, Keedy K, Fernandes P, Cohen-Wolkowiez M. Solithromycin Pharmacokinetics in Plasma and Dried Blood Spots and Safety in Adolescents. Antimicrob Agents Chemother. 2016 Mar 25;60(4):2572-6. doi: 10.1128/AAC.02561-15. Print 2016 Apr. PMID 26883693